CLINICAL TRIAL: NCT05576454
Title: A Randomized, Double-blinded, Single-dose, 3-arm Parallel Comparative Study on Pharmacokinetics and Safety of BAT2606 Injection Versus Mepolizumab Injection (EU-licensed Nucala® and US-licensed Nucala®) in Healthy Chinese Male Subjects
Brief Title: Evaluate the Pharmacokinetics of BAT2606 Injection in Healthy Chinese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BAT-2606-001-CR
Record Dates: First submitted 2022-10-08; First posted 2022-10-12 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-02

CONDITIONS: Severe Asthma
MeSH Terms: conditions — Asthma | interventions — mepolizumab

STUDY DESIGN:
Intervention Model Description: It's a randomized, double-blinded, single-dose, 3-arm parallel comparative study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blinded design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BAT2606 Injection (Experimental): PFS, Strength: 100 mg/1 mL, 100 mg, Subcutaneous injection.
  Interventions: Drug: Mepolizumab Injection (BAT2606 Injection)
- Mepolizumab Injection (EU-licensed Nucala®) (Active Comparator): PFS, Strength: 100 mg/1 mL, 100 mg, Subcutaneous injection.
  Interventions: Drug: Mepolizumab Injection (EU-licensed Nucala)
- Mepolizumab Injection (US-licensed Nucala®) (Active Comparator): PFS, Strength: 100 mg/1 mL, 100 mg, Subcutaneous injection.
  Interventions: Drug: Mepolizumab Injection (US-licensed Nucala)

INTERVENTIONS:
Drug: Mepolizumab Injection (BAT2606 Injection) — In this group, each subject will receive single subcutaneous injection of 100 mg BAT2606 Injection.
  Other Names: BAT2606 Injection
  Arms: BAT2606 Injection
Drug: Mepolizumab Injection (EU-licensed Nucala) — In this group, each subject will receive single subcutaneous injection of 100 mg Mepolizumab Injection (EU-licensed Nucala®).
  Other Names: EU-licensed Nucala
  Arms: Mepolizumab Injection (EU-licensed Nucala®)
Drug: Mepolizumab Injection (US-licensed Nucala) — In this group, each subject will receive single subcutaneous injection of 100 mg Mepolizumab Injection (US-licensed Nucala®).
  Other Names: US-licensed Nucala
  Arms: Mepolizumab Injection (US-licensed Nucala®)

SUMMARY:
To evaluate the pharmacokinetics, safety and immunogenicity of BAT2606 in healthy China male subjects.

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blind, single-dose, parallel three arms comparative study of pharmacokinetics, safety and immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects have signed the informed consent before the trial, and fully understood the content, process and relevant risks of the trial.
* 2. Subjects who are able to complete the study in accordance with the requirements of the protocol.
* 3. Visiting subjects (including partners) who are willing to comply with the study provisions agree to have no pregnancy plans and no donor sperm plans throughout the trial and for 6 months after dosing, and to voluntarily use effective contraception, as described in Appendix 4.
* 4. Subjects with BMI between 18 and 28 kg/m2 (both inclusive) and body weight between 55 and 85 kg (both inclusive).
* 5. Healthy Chinese male subjects between the ages of 18 and 55 years (both inclusive).
* 6. Subjects with normal or abnormal physical examinations without clinical significance.

Exclusion Criteria:

* 1. Subjects who have clinically significant abnormalities in clinical laboratory tests.
* 2. Subjects with clinical significance of abnormal ECG, chest x-ray.
* 3. Subjects with history of hypertension.
* 4. Subject who are or had been suffering from malignant neoplasm; subject who are or had been suffering from inflammatory bowel disease.
* 5. Subjects who have an active infection within 2 months prior to screening, including acute and chronic infections as well as localized infections.
* 6. Subjects who have active tuberculosis.
* 7. Subjects who have been exposed to TB within 3 months prior to screening.
* 8. Subjects whose T-cell test for tuberculosis infection (T-SPOT.TB) results are positive.
* 9. Subjects who are positive for HBsAg on the hepatitis B half test.
* 10. Subjects who have had a major injury or undergone previous surgical procedures or fracture within 4 weeks prior to enrollment.
* 11. Subjects who have taken any prescription medication within 28 days prior to screening.
* 12. Subjects who participate in another drug clinical trial within 3 months prior to enrollment.
* 13. Subjects who suffered an acute illness from the screening period until study drug administration.
* 14. Subjects who have received Mepolizumab (or its biosimilar) within 6 months (or within 5 half-lives of the drug, whichever is longer) prior to screening.
* 15. Subjects who have received live vaccination during the study period within 12 weeks prior to study dosing.
* 16. Subjects who are suspected or confirmed to be allergic (allergic to multiple medications or foods).
* 17. Subjects who smoked more than 5 cigarettes per day in the 3 months prior to screening.
* 18. Subjects who have taken any alcohol-containing product within 24h prior to study dosing.
* 19. Subjects who have donated blood or lost a significant amount of blood (> 450 mL) within 3 months prior to study drug administration.
* 20. Subjects with a positive urine drug screening.
* 21. Subject who is deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy Chinese male subjects between the ages of 18 and 55 years (both inclusive).
Enrollment: 207 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
Cmax | Day1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 15, 22, 29, 43, 57, 71, 85, 99, 113
  Maximum blood concentration
AUC0-∞ | Day1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 15, 22, 29, 43, 57, 71, 85, 99, 113
  Area under the plasma concentration-time curve from zero to infinity, AUC0-∞ = AUC0-t + Ct/λz

SECONDARY OUTCOMES:
AUC0-t | Day1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 15, 22, 29, 43, 57, 71, 85, 99, 113
  Area under the blood concentration-time curve from time 0 to the last time point at which the concentration can be measured
Tmax | Day1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 15, 22, 29, 43, 57, 71, 85, 99, 113
  Observed time to peak concentration
t1/2 | Day1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 15, 22, 29, 43, 57, 71, 85, 99, 113
  Elimination half-life t1/2 = 0.693/λz
CL/F | Day1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 15, 22, 29, 43, 57, 71, 85, 99, 113
  Total clearance rate, CL/F=Dose/AUC0-∞
Vd | Day1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 15, 22, 29, 43, 57, 71, 85, 99, 113
  Apparent volume of distribution, Vd =Dose/(AUC0-∞ × λz)
λz | Day1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 15, 22, 29, 43, 57, 71, 85, 99, 113
  Terminal elimination rate constant. The negative of the slope value obtained by taking the logarithm of the drug concentration and performing a linear regression against time is the terminal elimination rate constant
Adverse events | Day1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 15, 22, 29, 43, 57, 71, 85, 99, 113
  AE and SAE
Immunogenicity | Day1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 15, 22, 29, 43, 57, 71, 85, 99, 113
  Anti-drug antibody (ADA) positivity, ADA titer and neutralizing antibody (NAb) positivity for ADA.

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, PhD, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li C, Sun J, Xu J, Wu M, Li X, Liu Z, Dong Q, Sun Y, Ding Y. Comparison of pharmacokinetic similarity, immunogenicity, and safety of mepolizumab and BAT2606 in healthy Chinese men in a double-blinded, randomized, single-dose, three-arm parallel-group phase I trial. Front Pharmacol. 2025 Jul 25;16:1580883. doi: 10.3389/fphar.2025.1580883. eCollection 2025. PMID 40786037